CLINICAL TRIAL: NCT02902991
Title: The Study on the Clinical Utility of Liquid Biopsy in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Fei Ma, Department of Medical Oncology, National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing,China, Peking Union Medical College
Other Study IDs: CH-BC-052
Record Dates: First submitted 2016-09-04; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: liquid biopsy, breast cancer,circulating tumor biomarker
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumor cells,circulating tumor DNA and other liquid biopsy biomarkers

SUMMARY:
Through this prospective clinical trial,the investigators will focus on the relationship between circulating tumor biomarkers (i.e. circulating tumor cells, circulating tumor DNA and other biomarkers) and the status of primary tumor to discuss its application for assessing prognosis and individualized therapeutic direction. Moreover, the relationship between the circulating tumor cell subpopulations based on epithelial-mesenchymal transition and molecular pathological classification of breast cancer will be determined, which may enable the determination of the value of its application in therapeutic decision making.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years with histologically confirmed breast cancer.
* The patients diagnosed with breast cancer for the first time, including postoperative patients within one month and the patients diagnosed with Stage IV breast cancer for the first time.

Exclusion Criteria:

* The patients who has begun medication for breast cancer.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients diagnosed with breast cancer for the first time, including postoperative patients within one month and the patients diagnosed with Stage IV breast cancer for the first time.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
the enumeration of circulating tumor biomarkers | up to 2 years